CLINICAL TRIAL: NCT03455998
Title: Chronic Abdominal Pain After Gastric Bypass for Morbid Obesity
Brief Title: Chronic Abdominal Pain After Gastric Bypass
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Tom Mala, consultant, phd, Oslo University Hospital
Other Study IDs: Gastric bypass/pain
Record Dates: First submitted 2018-02-28; First posted 2018-03-07 (Actual); Last update posted 2018-03-13 (Actual); Status verified 2018-03

CONDITIONS: Abdominal Pain
Keywords: morbid obesity; gastric bypass; pain; symptoms
MeSH Terms: conditions — Abdominal Pain; Obesity, Morbid; Pain | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- post surgery: Patienst consultation Questionnaires
  Interventions: Other: questionnaires
- pre and post surgery: Patient consultation Questionnaires
  Interventions: Other: questionnaires

INTERVENTIONS:
Other: questionnaires

SUMMARY:
The study aims to explore patients perception of chronic abdominal pain after Roux en Y gastric bypass surgery for morbid obesity. The investigators aim to describe characteristics of symptoms of pain. Potential risk factors for developing abdominal pain post gastric bypass will be explored.

DETAILED DESCRIPTION:
This is a single-center, prospective, longitudinal, cohort study performed at the Department of Morbid Obesity and Bariatric Surgery, Oslo University Hospital. Patients undergoing gastric bypass are eligible for inclusion. The study is approved by the Regional Committee for Medical and Health Research Ethics (no.2013/1263), South-East health region. All participants provide written consent for study paennrollment.

The participants are asked to fill inn a set of questionnaires before and during follow-up after gastric bypass surgery. Symptom characteristics are explored and evaluated. Quality of life is included in the analyses. The main outcome is findings at 2 years post surgery, but the patients will be followed for 5 years.

The investigators also aim to evaluate by objective measures the patients perception of pain by temperature and skin pressure stimulants before and after surgery (2 years).

ELIGIBILITY:
Inclusion Criteria:

• Indication for gastric bypass surgery i.e. BMI > 40 kg/m2 or BMI > 35 kg/m2 and obesity related comorbidity following failed attempts of sustained weight loss

Exclusion Criteria:

* Other indications for gastric bypass surgery than obesity
* Previous bariatric surgery
* Other concomitant surgical procedures for abdominal pain such as cholecystectomy

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Patients planned for bariatric surgery (gastric bypass) at a single center
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2014-02-01 (Actual); Primary Completion 2015-06-30 (Actual); Study Completion 2020-10-31 (Estimated)

PRIMARY OUTCOMES:
Chronic abdominal pain 2 years post gastric bypass surgery | Patient follow up complete 2020
  questionnaire

SECONDARY OUTCOMES:
Quality of life | patient follow up complete 2020
  questionnaire
Objective evaluation of pain perception | baseline and 2 years
  skin sensors

CONTACTS AND LOCATIONS:
Overall Officials: Tom Mala, MD.phd, Principal Investigator — Oslo University Hospital
Locations (1):
- Oslo university Hopsital, Oslo, Norway

IPD SHARING:
Plan to Share IPD: No